CLINICAL TRIAL: NCT07055529
Title: Comparison of Efficacy and Safety Psoralen Combined With Ultraviolet A (PUVA) Vs Tofacitinib in the Treatment of Generalized Vitiligo.
Acronym: (PUVA)
Status: Not yet recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Hayat Abad Medical Complex, Peshawar (Other Government)
Responsible Party: Principal Investigator, Syeda Sana Zaman, Trainee Medical Officer, Hayat Abad Medical Complex, Peshawar
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MTI-HMC Peshawar
Record Dates: First submitted 2025-06-15; First posted 2025-07-09 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2025-06

CONDITIONS: Vitiligo, Generalized
MeSH Terms: conditions — Vitiligo

STUDY DESIGN:
Intervention Model Description: No additional details
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A in which the patient will recieve PUVA therapy (Other): The Study will have two groups and in this group patients will recieve Psoralen combined with UVA (PUVA) therapy
  Interventions: Drug: Group A recieving PUVA therapy
- Group B in which the patient will be given Tofacitinib 5mg (Other): This study will have two groups and this group will recieve tablet tofacitinib 5mg
  Interventions: Drug: Group B receiving Tablet Tofacitinib

INTERVENTIONS:
Drug: Group A recieving PUVA therapy — This group A will recieve PUVA therapy twice weekly for 6 months
  Other Names: Psoralen combined with Ultraviolet A
  Arms: Group A in which the patient will recieve PUVA therapy
Drug: Group B receiving Tablet Tofacitinib — This group will be given tablet Tofacitinib 5mg twice daily for 6 months
  Arms: Group B in which the patient will be given Tofacitinib 5mg

SUMMARY:
This study aims to compare the efficacy and safety of PUVA versus Tofacitinib in the treatment of generalized vitiligo. Given the high prevalence of vitiligo in Pakistan and the significant psychosocial impact on patients, particularly in Peshawar, this study will provide valuable insights into optimal treatment strategies.

DETAILED DESCRIPTION:
Vitiligo is a chronic skin condition that occurs due to the loss of melanocytes, which results in the loss of skin colour. Vitiligo seems to be a common disease. An estimated 0.5-2% of people in the world suffer from it.1 It affects the quality of life because of being visible and often being stigmatized.1 In a study appearing in the Journal of Pakistan Association of Dermatologists, researchers studied familial prevalence and association of vitiligo with other auto-immune diseases in Pakistan. The study found 22% of vitiligo patients had a positive family history, thus suggesting a genetic predisposition. 2 There are many treatment options of varying efficacy available for vitiligo. For many years, PUVA (oral Psoralen plus ultraviolet A) therapy has been used to treat generalized vitiligo. This therapy promotes the repigmentation of the skin by facilitating the migration and proliferation of melanocytes. PUVA therapy has been shown to produce repigmentation rates between 50-75% in responsive patients, particularly on the face and trunk.3 However, PUVA therapy needs close monitoring due to the risk of phototoxicity, gastrointestinal symptoms and longer-term risks of skin aging and carcinogenesis.4 Recent times have seen a rise in the use of new treatments such as Janus kinase (JAK) inhibitors like Tofacitinib for generalized vitiligo.5 Tofacitinib an oral JAK inhibitor, works through the modulation of the immune response believed to cause the autoimmune destruction of melanocytes. Clinical trials show Tofacitinib has repigmentation rates of 45-65%, and is better tolerated than conventional therapies such as PUVA.6 In the study "Tofacitinib to Treat Refractory Progressive Vitiligo: A Retrospective Case Series," 25 patients with refractory progressive vitiligo were treated with oral tofacitinib. Out of these 16 (64%) patients, the progression of disease ceased. Almost half of these patients observed this effect within one month. In addition 10 patients (40%) showed various degrees of repigmentation. The study pointed out that tofacitinib with phototherapy had a significant effect on repigmentation rate. General findings indicate that oral tofacitinib is probably effective for intractable progressive vitiligo.7 JAK inhibitors are potentially a safer and effective alternative treatment option for vitiligo patients.8 Although useful, there isn't much direct knowledge of PUVA versus Tofacitinib efficacy in the Pakistani population. Due to variations in genetic make-up, environmental conditions, and access to healthcare, the present study serves as a justification for carrying out such studies in order to determine the best treatment option for patients with generalized vitiligo.

The objective of this study is to compare the efficacy and safety of PUVA and Tofacitinib in generalized vitiligo. Because of the high frequency of vitiligo in Pakistan and the considerable psychosocial impact of the disease on the patients of Peshawar, the current study will yield useful information regarding the best course of action on treatments.

OBJECTIVE To compare the efficacy and safety of PUVA versus Tofacitinib in the treatment of generalized vitiligo.

Operational Definitions

Vitiligo

Vitiligo is defined as a chronic skin condition characterized by the development of depigmented patches due to the loss of pigment producing cells in the basal layer of epidermis (melanocytes). In this study, generalized vitiligo refers to widespread, symmetrical depigmentation affecting more than 10% of the body surface area, diagnosed clinically by a consultant dermatologist based on characteristic appearance and distribution of lesions.

Efficacy

Efficacy in this study will refer to the degree of repigmentation achieved, which will be measured using the Vitiligo Area Scoring Index (VASI) (Annex-1) to assess the percentage of repigmented skin in affected areas. A treatment will be deemed effective if it achieves at least 50% repigmentation in depigmented patches, as evaluated by VASI over a six-month period.

Safety

Safety means that the treatment has no major negative effects linked to it. In this study, safety will be determined by the incidence of side effects such as gastrointestinal symptoms, skin irritation, or system reaction that are related to the treatment. Safety data will be sourced from patient-reported outcome and clinical evaluations.

Null Hypothesis: There is no difference between the efficacy of Tofacitinib and PUVA in the treatment of generalized vitiligo.

Alternate Hypothesis There is difference between the efficacy of Tofacitinib and PUVA in the treatment of generalized vitiligo.

Materials and Methods

Study Design: Randomized Control Trial

Setting: Department of Dermatology, MTI-Hayatabad Medical Complex (HMC), Peshawar.

Duration of Study: Six months after approval of the synopsis.

Sample Size: My sample size is 64 patients (32 in each group) taking 75%3 proportion of efficacy of PUVA versus 45%5 proportion of efficacy of Tofacitinib with 80% power of test and 5% significance level on WHO sample size calculator.

Sampling Technique: Consecutive non-probability sampling.

Sample Selection:

Inclusion Criteria:

* Patients of either gender aged 18-60 years.
* Patients with generalized vitiligo (depigmentation affecting more than 10% of the body surface area).

Exclusion Criteria:

* People with localised vitiligo as these patients are given topical medication because depigmentation affects less than 10% of the body surface area.
* People who've had any allergic reactions from taking Psoralen or Tofacitinib will not be enrolled in the study to prevent adverse reactions that can harm the patient and affect assessment of its effectiveness.
* Pregnant or lactating women: Due to unknown effects on pregnancy and breastfeeding, Psoralen and Tofacitinib should not be taken as they may pose fetal and neonatal risks.
* Patients with severe systemic illnesses or those currently receiving other immunomodulatory treatments will not be recruited in order to reduce confounding factors that will affect the immune response.
* People who have used a topical agent or undergone UV therapy in the last three months so that any lasting effects of these treatments are avoided, this will allow clearer evaluation of the study drugs' effects on vitiligo repigmentation.
* Avoid including patients with any history of thromboembolic or other significant cardiovascular events. The use of Tofacitinib has been associated with a greater risk of thromboembolic events and may pose a risk to the safety of these patients.
* Patients with active or chronic infections(including TB or hepatitis). As Tofacitinib has immunosuppressive properties and including such patients might have aggravated infections.

Data Collection Procedure:

Study will begin after getting approval of Hospitals' Ethical Committee and CPSP Karachi. The patients presenting to the Skin Opd of our hospital will be assessed after taking written informed consent form (Annex-2). Upon enrollment, detailed demographic information such as age, gender, occupation status, and duration of disease will be collected for each patient.

A extensive clinical examination will be performed to assess the extent of vitiligo, with depigmentation percentage recorded based on body surface area affected. This initial evaluation will establish a baseline for further comparison.

Patients will then be randomized into two groups using block randomization. Group A will receive PUVA therapy session, administered twice weekly. Group B will receive oral Tofacitinib (5 mg) twice daily. The treatments will be carried out over a six-month period.

Follow-up visits will be scheduled every two months, during which the degree of repigmentation will be assessed by standardized tools, such as visual analogue scales and body surface area measurements. In addition to efficacy evaluation, any adverse events will be documented during each visit.

At the end of the six-month treatment period, a final assessment will be conducted to evaluate the overall percentage of repigmentation and document any adverse effects encountered during the trial. All the above information will be recorded on a predesigned proforma (Annex-3) attached to this synopsis.

Data Analysis Procedure:

The collected data will be analyzed using SPSS version 26. Numerical variables such as age, duration of vitiligo, percentage of repigmentation, and body surface area affected will be presented as mean+SD/Median (IQR) after checking normality of test using Shapiro Wilk Test. Categorical variables, including gender and occupation status will be expressed as frequencies and percentages. Chi-square tests will be applied to compare categorical variables such as gender, adverse effects and efficacy between the two groups. Data will be stratified with age and gender to see effect modifiers. Post stratification chi-square test or Fischer Exact test will be applied between both groups keeping p value < 0.05 as significance level. All results will be presented as tables or graphs.

ELIGIBILITY:
Inclusion Criteria:

* • Patients of either gender aged 18-60 years, diagnosed with generalized vitiligo (depigmentation affecting more than 10% of the body surface area).

  * Stable vitiligo (no new lesions or progression of existing lesions in the last three months).

Exclusion Criteria:

* Patients with a history of photosensitivity or allergies to Psoralen or Tofacitinib in order to prevent adverse reactions that could compromise patient safety and interfere with treatment efficacy assessment.
* Pregnant or lactating women in order to ensure fetal and neonatal safety, as the effects of Psoralen and Tofacitinib on pregnancy and breastfeeding are not well studied and could pose potential risks.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 64 (Estimated)
Dates: Start 2026-06-01 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Assesment of repigmentation | Six Months
  Efficacy in this study will refer to the degree of repigmentation achieved, which will be measured using the Vitiligo Area Scoring Index (VASI) (Annex-1) to assess the percentage of repigmented skin in affected areas. A treatment will be deemed effective if it achieves at least 50% repigmentation in depigmented patches, as evaluated by VASI over a six-month period.

CONTACTS AND LOCATIONS:
Locations (1):
- MTI-HMC Peshawar, Peshawar, Khyber Pukhtunkhwa, Pakistan